CLINICAL TRIAL: NCT01800526
Title: A Pilot Study of N-acetylcysteine in Patients With Sickle Cell Disease
Acronym: NACinSCD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bloodworks (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Barbara A. Konkle, M.D., Director, Clinical and Translational Research, Bloodworks
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117090
Record Dates: First submitted 2013-01-21; First posted 2013-02-27 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia
Keywords: Sickle Cell Disease; Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral N-acetylcysteine (NAC) (Experimental): Eligible subjects who did not participate in Intravenous NAC or subjects who are at least 4 weeks after participation in Intravenous NAC, will be given Oral NAC at a dose of 2400mg daily, in two equally divided doses, for 4 weeks. Subjects will have blood drawn prior to beginning the phase and weekly for 4 weeks. At each visit interim medical events and adverse events will be collected.
  Interventions: Drug: N-Acetylcysteine
- Intravenous N-acetylcysteine (NAC) (Experimental): For part 1, Eligible subjects who did not participate in Oral NAC or subjects at least 4 weeks after oral NAC will receive IV NAC 150 mg/kg over 8 hours. At least four weeks after the first infusion, the subject will receive IV NAC 300 mg/kg over 8 hours.
  For part 2, Eligible subjects with sickle cell disease and hospitalization for VOC within the past 2 years, who now present in VOC will be enrolled. Subjects will receive IV NAC 75 mg/kg over 1 hour every 6 hours for 5 days or discharge, whichever occurs earlier.
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine — Oral and Intravenous administration of NAC

SUMMARY:
Part 1: A pilot study in patients with homozygous S (HbSS) or hemoglobin S with beta zero thalassemia(HbS-βo thalassemia), with the aim of examining the effect of intravenous NAC treatment on plasma VWF parameters and measures of redox and RBC function.

Part 2: A pilot study in patients with sickle cell disease admitted to the hospital in vaso-occlusive crisis to determine the effects of NAC infusions on plasma VWF parameters and measures of redox and RBC function, and on measures of pain and hospital length of stay.

DETAILED DESCRIPTION:
Two primary processes dominate the complications associated with sickle cell disease (SCD): vasoocclusion and hemolysis. The plasma and vessel wall adhesive protein von Willebrand factor (VWF) is thought to be involved in both of these processes, so strategies aimed at reducing its secretion or reactivity, which could decrease complications in patients with SCD, are being tested.

Based on prior studies, N-acetylcysteine (NAC) treatment may decrease VWF activity in patients with SCD and may be a useful adjunctive treatment in this disorder.

Part 1 enrolls stable outpatients with homozygous S (HbSS) or hemoglobin S with beta zero thalassemia (HbS-βo thalassemia), with the aim of examining the effect of NAC treatment on VWF parameters, measures of oxidation and RBC fragments. Patients receive IV NAC first at 150 mg/kg over 8 hours and if tolerated, at a later date at 300 mg/kg over 8 hours in the University of Washington Clinical Research Center. Blood is collected for laboratory assessment. Subjects are later offered enrollment in an oral phase.

Part 2, patients with a history of vaso-occlusive crisis (VOC) are approached in the outpatient setting to discuss the study. When admitted for VOC, subjects receive NAC as an IV infusion75 mg/kg every 6 hours for up to 5 days. Blood for laboratory assays are collected each morning and pain assessment is performed prior to and following each NAC infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years of age
2. Diagnosis of homozygous sickle cell (SS) or S-beta thalassemia with at least two episodes of vaso-occlusive crises (VOC) requiring narcotics in each of the past 2 years. For part 2 can include hemoglobin SC disease.
3. For females of reproductive age, use of contraception and negative pregnancy test

Exclusion Criteria:

1. An additional hematologic diagnosis
2. Hemoglobin (Hgb) < 7gm/dL for part 1, < 6 gm/dL for part 2.
3. Asthma requiring medication
4. Liver function tests [alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (BilliT) > three times upper normal limit for Part 1.
5. Chronic transfusion therapy, or transfusion within 2 months of enrollment. For part 2 anticipated need for simple or exchange transfusion during hospitalization.
6. VOC requiring narcotic therapy within the prior week or requiring hospitalization with discharge < 2 weeks prior to study enrollment for Part 1, for part 2 admission for VOC within 30 days.
7. Pregnancy or nursing
8. Receiving another investigational drug
9. Known allergy to NAC
10. Per subject's physician not medically stable enough to participate
11. Taking nitroglycerin, carbamazepine, or phosphodiesterase 5 (PDE5) inhibitors
12. Abnormal baseline coagulation tests (> 1.5 times normal limits)
13. Platelets <150,000/microliter for Part 1.
14. For part 2, already enrolled in study twice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Laboratory measures of VWF activity | Part 1, Prior to during and following one day infusion or during oral administration; Part 2, daily during infusion and just following infusion completion
  To determine if NAC, given intravenously as a one day infusion, orally as an outpatient or during hospitalization for VOC has an effect on VWF level or function.

SECONDARY OUTCOMES:
Laboratory measures of red blood cell hemolysis and oxidation | Red blood cell (RBC) lab measures will be drawn prior to infusion, at the end of the infusion, 1 and 3 days following the end of the infusion, once a week during oral administration, and daily during hospitalization
  To determine effects of NAC treatment on laboratory markers of sickle cell disease by measuring a) lactate dehydrogenase (LDH) B) reticulocyte count, and c) percent dense cells and on oxidation by measuring RBC glutathione.
Adverse events during and following NAC administration | Adverse events will be measured from time of consent to completion of study, with particular attention to times around and during administration.
  To assess safety by evaluating subjects for adverse events during and at time points following administration.
Pain during VOC | Before and following each NAC infusion while hospitalized
  Pain will be measured using visual analog scale and numerical rating scale at study entry, and before and at completion of each infusion during hospitalization for VOC
Use of pain medications in morphine equivalents | Morphine equivalents for the hospitalization during which NAC was administered compared to past VOC admissions
  Data on morphine equivalents administered during the study hospitalization will be compared to those of past admissions.
Hospital length of stay (LOS) | Days of hospitalization during study compared to past hospitalizations for VOC
  LOS will be calculated by days of hospitalization when study drug is administered compared to past LOS for VOC admissions

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Konkle, M.D., Principal Investigator — Univ. of Washington/Bloodworks Northwest
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be published at end of study and data made available to outside investigators after results are published by investigators